CLINICAL TRIAL: NCT05055232
Title: An Open-label, Multicenter, Phase I Dose Escalation and Expansion Study of XZP-3621 in Chinese Patients With ALK or ROS1 Rearrangement Non-small Cell Lung Cancer
Brief Title: A Phase I Study of XZP-3621 in Chinese Patients With ALK or ROS1 Rearrangement Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3621-1001
Record Dates: First submitted 2021-09-14; First posted 2021-09-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2021-09

CONDITIONS: ROS1 Rearrangement Non-small Cell Lung Cancer; ALK Rearrangement Non-small Cell Lung Cancer
Keywords: XZP-3621; Dose escalation and expansion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XZP-3621 (Experimental): The first part is a dose-escalation design in patients with ALK/ROS1-positive solid tumor. The second part is an expansion in non-small cell lung Cancer (NSCLC) characterized by abnormalities in ALK expression.
  Interventions: Drug: XZP-3621

INTERVENTIONS:
Drug: XZP-3621 — tablets, dosage ranged from 50 mg to 600 mg, quaque die（QD）with the meal.

SUMMARY:
This is a multicenter, open-label, dose escalation, and expansion human clinical study to observe the safety, tolerability, pharmacokinetics, and pharmacodynamics of XZP-3621 in single and multiple oral administrations in advanced NSCLC subjects with ALK rearrangement or ROS1 rearrangement, and to initially explore the efficacy of XZP-3621.The study was divided into two parts: dose escalation and dose expansion.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose escalation, and expansion human clinical study to observe the safety, tolerability, pharmacokinetics, and pharmacodynamics of XZP-3621 in single and multiple oral administrations in advanced NSCLC subjects with ALK rearrangement or ROS1 rearrangement, and to initially explore the efficacy of XZP-3621.The study was divided into two parts: dose escalation and dose expansion.

Dose escalation part:

The purpose of this section was to determine MTD and RP2D doses in advanced NSCLC subjects with ALK rearrangement or ROS1 rearrangement detected in tumor tissue samples or blood samples (test method is not limited).The safety and PK of single dose in human subjects in each group were first studied. After PK blood sample was collected 72 hours after single dose on day 1, continuous dose was administered once a day for 4 weeks to confirm the safety and pharmacokinetic characteristics of single dose and continuous dose.

In this study, Modified Fibonacci method was used for dose escalation. One subject was enrolled at the initial dose of 50mg. After that, according to the "3+3" dose escalation principle, the dose of 100mg (100%), 200mg (100%), 300mg (50%), 400mg (33%), 500mg (25%), 600mg (20%)and so on was incremented successively. Starting from the 100mg Qd dose group, 3 NSCLC subjects with ALK rearrangement or ROS1 rearrangement should be included per dose.If less than 3 NSCLC subjects were ALK rearrangement in any dose group due to inclusion of ROS1, and no ≥1 PR was observed in this group, additional ALK rearrangement NSCLC subjects should be added until the requirements are met. However, as long as the number of subjects in the corresponding dose group who have completed DLT observations meets the "3+3" principle of escalation, the addition of subjects to the ALK rearrangement should not affect the normal escalation of the next dose group.

Dose expansion part:

In the dose escalation study, if 2 out of 3 ALK rearrangement NSCLC subjects have a partial response (PR) or complete response (CR) after all subjects in the dose escalation study have completed DLT evaluation and confirmed that the dose is safe, that is, a dose extension study is performed from this dose to the MTD dose group. Each dose was reenrolled in about 15 NSCLC subjects with ALK rearrangement or ROS1 rearrangement demonstrated by Ventana immunohistochemistry or FISH or RT-PCR.

Subjects were treated with XZP-3621 for a 28-day treatment cycle, with continuous administration of or XZP-3621 until disease progression occurs, or an intolerable toxic reaction impeding further treatment occurs, or the investigator determines that the subject's current condition is unsuitable for further treatment, the informed consent is withdrawn, or the subject dies. RECIST efficacy was evaluated once every two treatment cycles.

During treatment, dose adjustments (both up and down) can be made according to protocol based on subjects' tolerance and the occurrence of adverse events related to the study drug. Only one dose reduction of the study drug is permitted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-75 years (including 18 and 75 years);
2. Stage IV NSCLC or Stage IIIB and IIIC NSCLC that cannot be treated with radical radiotherapy(IASLC); Dose escalation: ALK rearrangement or ROS1 rearrangement positive, the test specimen and method is not limited;Patients were required to have experienced treatment failure or disease progression after prior ALK inhibitor therapy or were unable to afford ALK inhibitors, regardless of other previous anti-tumor therapies.

   Dose expansion: ALK rearrangement or ROS1 rearrangement was confirmed by nationally approved Ventana immunohistochemistry or FISH or RT-PCR. There is no restriction on the number and type of antitumor therapy previously received; There is no limit to test time, test unit/kit and test specimen; Prior treatment was not limited, regardless of prior treatment with or without other antitumor therapy.
3. Dose escalation: ECOG score 0-1; Dose expansion: ECOG score 0-2;
4. Dose expansion: Subjects must have at least one measurable target lesion as defined by RECIST V1.1 and the lesion has not previously been treated with radiation or has had significant disease progression after radiation therapy;
5. All acute toxicities from prior anti-cancer treatment or complications/sequelae from surgical procedures are resolved to baseline or ≤ grade 1 (CTCAE V5.0, hair loss or other toxicities deemed by the investigator to pose no safety risk to the subject);
6. All previous antitumor therapies (including chemotherapy, radiotherapy and immunotherapy) have been stopped for at least 4 weeks before the first administration of XZP-3621 (in which nitrosoreas or mitomycin should be stopped for≥ 6 weeks, and oral small molecule targeted therapy drugs and Chinese medicine (including decoction or Chinese patent medicine) should be stopped for at least 2 weeks);Palliative radiation therapy (irradiation of non-target lesions, local administration of non-target lesions) for the purpose of relieving local symptoms was allowed to be completed one week before study enrollment;
7. The expected survival was determined by the investigator to be 12 weeks or more;
8. At the time of enrollment, the subject's organ function at baseline was good, and the laboratory data met the following criteria:

   1. Blood routine: Absolute Neutrophils Count≥1.5*109/L、PLT≥90*109/L、HGB≥90g/L;
   2. Liver function: Serum total bilirubin ≤1.5 * ULN；ALT and AST≤3 * ULN；ALT and AST ≤5*ULN (Liver metastases subjects);
   3. Renal function: CrCl≥50 mL/min /1.73 m2（≥0.835mL/s, according to Cockcroft-Gault formula;
   4. AMS≤ULN (If AMS is elevated, between 1 and 2 times of ULN, but there are no other signs and clinical evidence of pancreatic disease, the subject can be included);
   5. HbA1c≤ 7.0%;
9. The fertile male or female subject must agree to use an effective contraceptive method, such as a double-screen contraceptive method, a condom, oral or injectable contraceptive, an intrauterine device, etc. during the study period and within 90 days of the last dose of XZP-3621.
10. The subject has fully understood the study and signed the informed consent voluntarily.

Exclusion Criteria:

1. Subjects with primary CNS tumors or symptoms of brain metastases (except those with treated or untreated asymptomatic CNS metastases who had not been treated with corticosteroids for 2 weeks prior to enrollment, stereotactic radiotherapy for 1 week, and whole brain radiotherapy for 2 weeks prior to enrollment);
2. subject with small cell lung cancer;
3. Malignant thoracic cavity/peritoneal cavity effusion and/or pericardial effusion that cannot be controlled in the dose extension study;
4. Prior diagnosis of any other malignancy within 3 years prior to enrollment except for adequately treated and stable basal cell carcinoma or squamous skin cell carcinoma or carcinoma in situ of the cervix;
5. Subject has history of hematopoietic stem cell or bone marrow transplantation;
6. Subject has history of pancreatitis;
7. A history of cerebrovascular accident, including transient ischemic attack or stroke, within 6 months prior to enrollment;
8. Major surgery (defined as surgery under general anesthesia or surgery with significant incisions) or unresolved postoperative complications prior to administration of XZP-3621 within 4 weeks prior to enrollment;
9. Chronic Hepatitis B(HBV), or/and HBV DNA>500 IU/ml, Hepatitis C(HCV);
10. known human immunodeficiency virus (HIV);
11. Body temperature is above 37.5℃ or significant active infections that can influence the clinical study, including active tuberculosis;
12. Uncontrollable electrolyte disturbances, such as low calcium, low magnesium, and low kalemia, may affect the elongation of QTc;
13. Unable to swallow;
14. History of large area diffusion/double pulmonary fibrosis, or known grade 3 or 4 pulmonary fibrosis, or current with clinically significant active pulmonary diseases, including pneumonia, allergic pneumonia, interstitial pneumonia and other interstitial lung diseases, and bronchiolitis oblationus, currently suffering from radiation pneumonia requiring hormone therapy, but not includ a history of previous radiation pneumonia;
15. Subjects with impaired heart function or clinically significant heart disease;
16. Clinically significant gastrointestinal abnormalities, including active ulcerative colitis, chronic diarrhea due to intestinal malabsorption, Crohn's disease, and/or prior surgery affecting absorption;
17. Any serious and/or uncontrolled comordities that the investigator believes may interfere with the study assessment, such as uncontrolled hypertension (defined as systolic blood pressure ≥140mmHg and/or diastolic blood pressure ≥90mmHg at rest) and clinically significant neurological disorders;
18. Subjects are receiving drugs known to strongly inhibit or induce CYP3A4 and should not stop taking them one week before administration XZP-3621 and during the study period (or within the five half-lives of the drug, whichever is longer);
19. The subject is scheduled for surgery, or the investigator determines that the subject needs surgery;
20. Participation in any other clinical trial within 1 month prior to enrollment (except those who had been removed from other clinical studies and only had survival follow-up);
21. Allergic constitution or a history of severe allergies;
22. Pregnant women and breastfeeding women;
23. Other conditions that the investigator considered unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events/serious adverse events | From screening stage to 30 days after study completion.
  Characterization of the safety and tolerability of XZP-3621 as determined by changes in laboratory values and electrocardiograms
Incidence rate of dose limiting toxicities (DLTs) during the first cycle of treatment | 4 weeks
  Maximum Tolerated Dose(s) (MTD(s)) and/or recommended phase 2 dose (RP2D(s)) of XZP-3621 in ALK-positive non-small cell lung cancer (NSCLC) patients. Cycle = 4 weeks.
Maximum tolerated dose（MTD） | 4 weeks
  The MTD is determined by the number of the participants in cohort who suffer a dose-limiting toxicity (DLT). The MTD is defined as the former dose at which more than one third of the participants develop a DLT. If no DLTs are observed, the MTD is not reached.

SECONDARY OUTCOMES:
Objective response rate(ORR) | 8 weeks
  Imaging assessments were performed every 2 treatment cycles until tumor progression/recurrence. It was defined as the proportion of patients evaluated as having complete response (CR) or partial response (PR) according to RECIST1.1 criteria
Duration of response(DoR) | 8 weeks
  For subjects with CR or PR only, defined as the time from the date of first remission to the date of disease progression (PD) or death.
Progress free survival(PFS) | 8 weeks
  It was defined as the time from the first study drug treatment to disease progression or death.
Cmax | 4 weeks
  Pharmacokinetics of XZP-3621 by assessment of maximum plasma XZP-3621 concentration.
Tmax | 4 weeks
  Pharmacokinetics of XZP-3621 by assessment of time to Cmax.

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD, Principal Investigator — Shanghai Chest hospital affiliated to Shanghai jiao tong university
Locations (1):
- Shanghai Chest hospital affiliated to Shanghai jiao tong university, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ai X, Guo R, Zhang L, Fang J, Zhang Y, Chen J, Zhao J, Ye F, Wang S, Shi M, Zhang X, Zhang F, Li J, Wang L, Guo X, Xu L, Duan X, Hu Y, Lu S. Preclinical characterization and first-in-human, phase I trial of the novel ALK inhibitor dirozalkib in advanced non-small cell lung cancer. Eur J Cancer. 2026 Jan 7;235:116221. doi: 10.1016/j.ejca.2026.116221. Online ahead of print. PMID 41539180